CLINICAL TRIAL: NCT07091305
Title: A Study of QL1706 Combined With Chemotherapy Induction on Sequential Immunotherapy Consolidation in Patients With Limited-Stage Small Cell Lung Cancer After Chemoradiotherapy：A Phase II Trial
Brief Title: A Study of QL1706 Combined With Chemotherapy Induction on Sequential Immunotherapy Consolidation in Patients With Limited-Stage Small Cell Lung Cancer After Chemoradiotherapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xuwei Cai, Director, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IS25129
Record Dates: First submitted 2025-07-02; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Limited-stage Small Cell Lung Cancer (LS-SCLC); Chemoradiotherapy; Induction Therapy; Consolidation Immunotherapy
Keywords: Limited-stage small cell lung cancer; QL1706; chemoradiotherapy; induction therapy; consolidation immunotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Induction: QL1706 combined with Etoposide and platinum, intravenous infusion (IV), every 3 weeks.
  Chemoradiotherapy, followed by QL1706 consolidation, intravenous infusion (IV), every 3 weeks.
  Interventions: Drug: QL1706 (bispecific antibody targeting PD-1 and CLTA-4)

INTERVENTIONS:
Drug: QL1706 (bispecific antibody targeting PD-1 and CLTA-4) — Induction: QL1706 5 mg/kg IV on Day 1, Etoposide: 100 mg/m² IV on Days 1-3, Cisplatin or Carboplatin: Cisplatin 75 mg/m² IV on Day 1 or Cisplatin 25 mg/m² IV on Days 1-3, Or Carboplatin AUC = 5 IV on Day 1, Q3W, for a total of 2 cycles.
  Chemoradiotherapy：Thoracic Radiotherapy（60 Gy in 30 fractions, once daily (2 Gy/fraction), or 45 Gy in 30 fractions, twice daily (1.5 Gy/fraction)），Etoposide 100 mg/m² IV on Days 1-3, Cisplatin either 75 mg/m² IV on Day 1, or 25 mg/m² IV on Days 1-3, Or Carboplatin AUC=5 IV on Day 1 PCI: Patients achieving or approaching complete response, per investigator assessment, 25Gy in 10 fractions.
  Consolidation: QL1706 5 mg/kg IV on Day 1, Q3W

SUMMARY:
The study is being conducted to evaluation of the Efficacy and Safety of QL1706 Combined with Chemotherapy Induction in Sequential Immunotherapy Consolidation After Concurrent Chemoradiotherapy for Limited-Stage Small Cell Lung Cancer(LS-SCLC), and Exploration of the Correlation Between Biomarkers (PD-L1, TMB, ctDNA, etc.) Related to QL1706 Treatment and Treatment Efficacy and Prognosis.

QL1706 (Iparomlimab and Tuvonralimab) is a single bifunctional MabPair product against PD-1 and CTLA-4. QL1604 is a monoclonal antibody against PD-1.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be aged between 18 and 75 years (inclusive of boundary values), and both males and females are eligible.
2. Pathologically confirmed LS-SCLC
3. Investigator confirmation of at least one measurable lesion, as defined by RECIST v1.1
4. ECOG performance status of 0 or 1
5. Forced expiratory volume in one second (FEV₁) > 1.0 L
6. No clinically significant interstitial lung disease on baseline CT or PET/CT.
7. Adequate organ and bone-marrow function (all tests performed within 7 days prior to first dose; no transfusions, growth factors, albumin, or other corrective therapies within 14 days):Hemoglobin ≥ 90 g/L, ANC ≥ 1.5 × 10⁹/L, PLT ≥ 90 × 10⁹/L,Serum creatinine ≤ 1.5 × ULN, TBIL ≤ 1.5 × ULN, ALT and AST ≤ 3 × ULN, Albumin (ALB) ≥ 25 g/L,INR ≤ 1.5 × ULN, PT and APTT ≤ 1.5 × ULN (subjects on prophylactic anticoagulation must have values within a safe therapeutic range, per investigator)
8. Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to enrollment and agree to use reliable contraception from screening until 3 months after the last dose; male subjects must agree to use effective contraception or have undergone surgical sterilization for the same period.
9. No prior systemic anti-tumor therapy before enrollment.
10. Estimated life expectancy ≥ 12 weeks.

Exclusion Criteria:

1. Known hypersensitivity to QL1706 or any of its excipients
2. Histologically confirmed non-small cell lung cancer (NSCLC) or mixed tumor containing an NSCLC component.
3. History of another primary malignancy or previous allogeneic organ transplantation.
4. Surgery (other than diagnostic biopsy) within 4 weeks before first dose of study drug.
5. Active substance abuse (e.g., illicit drug use), chronic alcoholism, AIDS, or known HIV infection.
6. Active autoimmune disease, or history of autoimmune disease likely to recur. Systemic corticosteroid therapy equivalent to >10 mg/day prednisone (or other immunosuppressive therapies) within 14 days before first dose.
7. Prior therapy with any antibody or agent targeting T-cell co-regulatory proteins (e.g., PD-1, PD-L1, CTLA-4, TIM-3, LAG-3).
8. Interstitial lung disease (ILD), or history of ILD requiring steroid therapy. History of idiopathic pulmonary fibrosis, drug-induced pneumonitis, organizing pneumonia (e.g., bronchiolitis obliterans), or evidence of active pneumonia on screening chest CT.
9. Live vaccine administration within 28 days prior to first study drug dose. Any condition or comorbidity contraindicating chemo- or radiotherapy (e.g., active infection, myocardial infarction within 6 months, symptomatic heart disease including unstable angina, congestive heart failure, uncontrolled arrhythmia, ongoing immunosuppressive therapy).
10. Pregnant or breastfeeding women; women of childbearing potential or men unwilling to use adequate contraception.
11. Known hereditary bleeding diathesis or coagulation disorder.
12. Prior malignancy, except adequately treated non-melanoma skin cancer, or in situ carcinoma (e.g., breast, oral, cervical) with expected survival >3 years.
13. Any other medical, psychiatric, or laboratory abnormality that, in the investigator's judgment, could interfere with trial participation or interpretation of results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 12 months after the last participant entry
  To evaluate the efficacy of QL1706 combined with chemotherapy as induction therapy followed by chemoradiotherapy (CRT) for patients with LS-SCLC as measured by investigator-assessed PFS

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 12 months after the last participant entry
  To evaluate the efficacy of QL1706 combined with chemotherapy as induction therapy followed by chemoradiotherapy (CRT) for patients with LS-SCLC as measured by investigator-assessed OS
Objective Response Rate (ORR) | through study completion, an average of 12 months after last patient entry
  Assessed according to RECIST V1.1.The Objective Response Rate (ORR) is defined as the best ORR during the study period, including cases of Complete Response (CR) and Partial Response (PR)
Duration of Response (DoR) | time from the first tumor assessment showing response to disease progression or death (whichever occurs first),assessed up to 24 months
  For patients who achieve Complete Response (CR) or Partial Response (PR), the time from the first tumor assessment showing response to disease progression or death (whichever occurs first).
Disease Control Rate (DCR) | through study completion, an average of 12 months
  DCR refers to the percentage of cases with the best efficacy evaluation of "Complete Response (CR) + Partial Response (PR) + Stable Disease (SD)
Quality-of-life(QoL) | Through study completion, an average of 12 months after last participant entry
  QoL scores will be transformed to a scale of 0-100 according to the EORTC QLQ scoring manual. Mean scores will be compared at each assessment timepoint, and a difference of 10 points is considered clinically relevant.
Correlation between outcomes of study treatment and biomarkers in tissue, blood | Through study completion, an average of 2 years after last patient entry
  A detailed plan for analyses will be defined when sufficient material for translational research has been collected.
Adverse events(AE) | through study completion, an average of 12 months
  Number of participant with treatment-related adverse events assessed based on CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No